CLINICAL TRIAL: NCT04962308
Title: An Open-label,Phase Ⅳ Clinical Trial to Evaluate the Immunogenicity and Safety of the Inactivated SARS-CoV-2 Vaccine (Vero Cell) in Healthy Population Aged From 18 to 59 Years.
Brief Title: Clinical Trial of Inactivated SARS-CoV-2 Vaccine for Prevention of COVID-19 in Healthy Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-4003
Record Dates: First submitted 2021-07-13; First posted 2021-07-14 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): 200 subjects in group A1 will receive one dose of booster immunization 3 months after the completion of the second dose of primary immunization of the SARS-CoV-2 Inactivated vaccine.
  Interventions: Biological: SARS-CoV-2 Inactivated Vaccine
- Control Group (Experimental): 200 subjects in group A2 will receive one dose of booster immunization 5 months after the completion of the second dose of primary immunization of the SARS-CoV-2 Inactivated vaccine.
  Interventions: Biological: The SARS-CoV-2 Inactivated Vaccine
- Safety group (Experimental): 1000 subjects in group B will be enrolled and receive 1 dose of booster immunization more than 3 months after the completion of the second dose of primary immunization of the SARS-CoV-2 Inactivated vaccine
  Interventions: Biological: SARS-CoV-2 Inactivated Vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 Inactivated Vaccine — 600SU inactivated virus in 0·5 mL of aluminiumhydroxide solution per injection
  Other Names: CoronaVac
  Arms: Experimental Group; Safety group
Biological: The SARS-CoV-2 Inactivated Vaccine — 600SU inactivated virus in 0·5 mL of aluminiumhydroxide solution per injection
  Other Names: CoronaVac
  Arms: Control Group

SUMMARY:
This study is an open-label phase Ⅳ clinical trial of the inactivated SARS-CoV-2 vaccine(CoronaVac)manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the immunogenicity and safety of the Inactivated SARS-CoV-2 Vaccine (Vero Cell) in Healthy Population Aged From 18 to 59 Years.

DETAILED DESCRIPTION:
This study is an open-label phase Ⅳ clinical trial in healthy adult aged 18-59 years. The experimental vaccine was manufactured by Sinovac Research and Development Co.,Ltd.. A total of 1400 subjects will be enrolled,the safety and immunogenicity of booster immunization were evaluated in 400 subjects (group A) who received two doses of primary immunization at an interval of 21 to 31 days. And the safety of booster immunization was evaluated in the extended safety group (group B), which included 1000 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-59;
* Have been received two doses of inactivated SARS-CoV-2 vaccine(CoronaVac)manufactured by Sinovac Research & Development Co., Ltd at an interval of 21 to 31 days for group A.Have been vaccination two doses of inactivated SARS-CoV-2 vaccine(CoronaVac)manufactured by Sinovac Research & Development Co., Ltd for group B;
* The subjects can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* History of SARS-CoV-2 infection;
* Any serious adverse reactions that are causally related to vaccination during the primary immunization of the previous inactivated SARS-CoV-2 vaccine;
* Severe allergic reactions after primary immunization (including urticaria/rash within 30 minutes after vaccination);
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) within 6 months before primary immunization and before booster immunization;
* Already pregnant or are breastfeeding, planning to get pregnant (according to subjects' self-report and urine pregnancy test results)
* Receipt of attenuated live vaccines within 14 days prior to booster vaccination;
* Receipt of inactivated or subunit vaccines within 7 days prior to booster vaccination;
* Acute diseases or acute exacerbation of chronic diseases within 7 days prior to booster vaccination;
* Axillary temperature >37.0°C prior to booster vaccination;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1400 (Estimated)
Dates: Start 2021-06-19 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-12-19 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer(GMT) of neutralizing antibody to live SARS-CoV-2 | 1 month after booster immunization
  GMT of the neutralizing antibody to live SARS-CoV-2 within 1month after booster immunization of the Inactivated SARS-CoV-2 vaccine.
Safety index-incidence of adverse reactions | 1 month after booster immunization
  Incidence rate of adverse reactions within 1 month after booster immunization of the Inactivated SARS-CoV-2 vaccine

SECONDARY OUTCOMES:
Safety index-incidence of serious adverse events | 1 month after booster immunization
  Incidence rate of serious adverse events within 1 month after booster immunization of the Inactivated SARS-CoV-2 vaccine
Seroconversion rate,seropositivity rate and GMI of the neutralizing antibody to SARS-CoV-2 | 1 month after booster immunization
  Seroconversion rate,seropositivity rate and GMI of the neutralizing antibody to SARS-CoV-2 within 1 month after booster immunization of the Inactivated SARS-CoV-2 vaccine
Seropositivity rate of IgG antibody | 1 month after booster immunization
  Seropositivity rate of IgG antibody within 1 month after booster immunization of the Inactivated SARS-CoV-2 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Master, Principal Investigator — Beijing Center for Disease Control and Prevention
Locations (1):
- Beijing Centers for Diseases Control and Prevention, Beijing, China